CLINICAL TRIAL: NCT00032617
Title: CSP #494 - A Randomized Clinical Trial of Cognitive-Behavioral Treatment for PTSD in Women (PTSD)
Brief Title: A Randomized Clinical Trial of Cognitive-Behavioral Treatment for Post-Traumatic Stress Disorders in Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Friedman, Matthew - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 494
Record Dates: First submitted 2002-03-27; First posted 2002-03-28 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Stress Disorder; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress Disorders, Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Prolonged Exposure
  Interventions: Procedure: Prolonged Exposure
- 2 (Active Comparator): Present Centered Therapy
  Interventions: Procedure: Present Centered Therapy

INTERVENTIONS:
Procedure: Prolonged Exposure — trauma-focused exposure therapy
  Arms: 1
Procedure: Present Centered Therapy — therapy that focuses on current problems
  Arms: 2

SUMMARY:
The purpose of the proposed DVA cooperative study is to evaluate the efficacy of exposure therapy for treating PTSD and associated problems in female veterans and active duty military personnel. We propose to compare exposure therapy, Prolonged Exposure, with a comparison therapy that focuses on current problems, Present Centered Therapy.

The study is a randomized clinical trial involving 384 female veterans and active duty personnel in 11 VA medical centers and 1 DoD medical center. All subjects, even self-referrals, will enter the study through referrals by mental health clinicians at the participating sites. Following informed consent, subjects will be screened for inclusion and exclusion diagnoses. If they meet these criteria and agree to participate, they will be randomly assigned to one of the two treatments, which will occur weekly for 10 weeks. Subjects will be assessed before treatment, immediately following treatment, and 3 and 6 months after the end of treatment. The primary outcome is PTSD severity. Secondary outcomes are anxiety and depression. Exploratory outcomes include associated features of PTSD, such as dissociation and substance abuse; psychosocial functioning, quality of life, physical health, satisfaction with treatment, and service utilization. Both treatments will be described in detail in a treatment manual and monitored intensively to ensure that they are administered correctly.

DETAILED DESCRIPTION:
Intervention: Patients will be randomized to one of two interventions: Prolonged Exposure (PE) consisting of 10 weekly treatment sessions that include education about and exposure to the memories of the trauma to which the patient was engaged; or Present Center Therapy (PCT), which will consist of a control therapy of the same duration that will provide emotional support for the trauma victim.

Primary Hypothesis: Prolonged Exposure (PE) will be more effective than Present-Centered Therapy (PCT) for the treatment of PTSD due to military-related trauma in women veterans. PE specifically targets PTSD symptoms, and the CAPS, our primary outcome measure. The Clinician Administered PTSD Scale (CAPS) is considered to be the gold-standard for PTSD assessment.

Secondary Hypothesis: PE will be more effective than PCT for treating the anxiety and depression that often are comorbid with PTSD.

Study Abstract: As noted in a recent report on the VA Women's Health Project, it is important to study women veterans because they are increasingly seeking VA health care. For many women veterans, Posttraumatic Stress Disorder (PTSD) is a specific healthcare concern that is associated with substantial psychosocial and functional disability.

The study was proposed in response to the Research Priority Announcement on Posttraumatic Stress Disorder research issued August 1, 1997, as a study aimed a special subpopulation of VA patients with PTSD: women veterans who have been traumatized during their military service.

The first planning meeting for the study was held January 20-21, 2000 in Washington, DC. The protocol was submitted on August 1, 2000; it was reviewed and approved by the Cooperative Studies Evaluation Committee on October 10, 2000. Intake of training cases is expected to begin 01/01/2002.

ELIGIBILITY:
Inclusion Criteria:

* female veterans or active duty personnel with a current diagnosis of PTSD due to any type of trauma;
* have experienced trauma no less than 3 months prior to entering the trial;
* have at least one clear memory of the trauma that caused their PTSD (sufficient for constructing a scene to be used in PE);
* consent to be randomized into treatment;
* not receive other psychotherapy for PTSD during the 10 weeks of active treatment;
* psychotherapy for other problems, brief check-ins with an existing therapist, and attendance at self-help groups will be allowed;
* if on psychoactive medication be on a stable medication regimen for a minimum of 2 months prior to entering the trial.

Exclusion Criteria:

* current substance dependence;
* prior substance dependence that has not been in remission at least 3 months;
* any current psychotic symptoms; current Mania or Bipolar Disorder;
* prominent current suicidal or homicidal ideation;
* any severe cognitive impairment or history of Organic Mental Disorder;
* current involvement in a violent relationship;
* self-mutilation within the past 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2002-08; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
summing totals of 17 DSM-IV symptoms | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Friedman, MD PhD, Study Chair — VA Medical & Regional Office Center
Locations (13):
- United States (13):
  - VA Eastern Colorado Health Care System, Denver, Denver, Colorado
  - VA Medical Center, Bay Pines, Bay Pines, Florida
  - Atlanta VA Medical and Rehab Center, Decatur, Decatur, Georgia
  - Southeast Veterans Healthcare System, New Orleans, New Orleans, Louisiana
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - Walter Reed (DCI-HUC), Bethesda, Maryland
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - New Mexico VA Health Care System, Albuquerque, Albuquerque, New Mexico
  - VA Medical Center, Cincinnati, Cincinnati, Ohio
  - VA Medical Center, Cleveland, Cleveland, Ohio
  - VA Medical Center, Portland, Portland, Oregon
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - VA Medical & Regional Office Center, White River Junction, Vermont

REFERENCES:
- [Derived] Stirman SW, Cohen ZD, Lunney CA, DeRubeis RJ, Wiley JF, Schnurr PP. A personalized index to inform selection of a trauma-focused or non-trauma-focused treatment for PTSD. Behav Res Ther. 2021 Jul;142:103872. doi: 10.1016/j.brat.2021.103872. Epub 2021 Apr 26. PMID 34051626
- [Derived] Schnurr PP, Lunney CA. Residual symptoms following prolonged exposure and present-centered therapy for PTSD in female veterans and soldiers. Depress Anxiety. 2019 Feb;36(2):162-169. doi: 10.1002/da.22871. Epub 2018 Dec 21. PMID 30576030
- [Derived] Lunney CA, Schnurr PP, Cook JM. Comparison of clinician- and self-assessments of posttraumatic stress symptoms in older versus younger veterans. J Trauma Stress. 2014 Apr;27(2):144-51. doi: 10.1002/jts.21908. Epub 2014 Apr 2. PMID 24700623
- [Derived] Rosen CS, Greenbaum MA, Schnurr PP, Holmes TH, Brennan PL, Friedman MJ. Do benzodiazepines reduce the effectiveness of exposure therapy for posttraumatic stress disorder? J Clin Psychiatry. 2013 Dec;74(12):1241-8. doi: 10.4088/JCP.13m08592. PMID 24434093
- [Derived] Wolf EJ, Lunney CA, Miller MW, Resick PA, Friedman MJ, Schnurr PP. The dissociative subtype of PTSD: a replication and extension. Depress Anxiety. 2012 Aug;29(8):679-88. doi: 10.1002/da.21946. Epub 2012 May 25. PMID 22639402
- [Derived] Schnurr PP, Friedman MJ, Engel CC, Foa EB, Shea MT, Chow BK, Resick PA, Thurston V, Orsillo SM, Haug R, Turner C, Bernardy N. Cognitive behavioral therapy for posttraumatic stress disorder in women: a randomized controlled trial. JAMA. 2007 Feb 28;297(8):820-30. doi: 10.1001/jama.297.8.820. PMID 17327524